CLINICAL TRIAL: NCT06333054
Title: A Randomised, Controlled, Investigator Blinded, Comparative Study to Evaluate the Safety and Efficacy of a Head Lice Shampoo.
Brief Title: Safety and Efficacy of a Head Lice Shampoo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oystershell NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCLIN0091/ 14ct/mp37li
Record Dates: First submitted 2024-03-19; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Head Lice

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Silcap Shampoo (Experimental): Subjects with head lice were treated with Silcap Shampoo at visit 1 (day 0) and at visit 3 (day 7).
  Interventions: Device: Silcap Shampoo
- Goldgeist® Forte (Active Comparator): Subjects with head lice were treated with Goldgeist® Forte at visit 1 (day 0) and at visit 3 (day 7).
  Interventions: Drug: Pyrethrum Extract

INTERVENTIONS:
Drug: Pyrethrum Extract — Treatment with Goldgeist® Forte
  Arms: Goldgeist® Forte
Device: Silcap Shampoo — Treatment with Silcap Shampoo
  Other Names: Paranix
  Arms: Silcap Shampoo

SUMMARY:
This study is designed to compare the effectiveness and safety of test head lice shampoo (Test product) versus Goldgeist® Forte (reference product) following two applications.

DETAILED DESCRIPTION:
The primary objective was to show, that the cure rate after local application of Test head lice shampoo is better than a predefined limit. It had to be shown, that the Test head lice shampoo achieved a cure rate superior to 70% (cure rate at the end of day 10, corrected for re-infestation).

ELIGIBILITY:
Inclusion Criteria:

* Gender: male/female
* Age: ≥ 1 year of age at the time of signing the informed consent
* Patients with active head lice infestation of at least 5 living lice and 5 apparently living eggs
* Patient or his/her guardian must be capable of understanding and providing written informed consent
* The patient or his/her legal representative must give written informed consent, after having been oral and written informed about benefits and potential risks of the trial, as well as details of the insurance taken out to cover the subjects participating in the study
* Patients must agree to not use any other ant-lice treatment for the duration of the study
* Female patients:

are women of childbearing potential who test negative for pregnancy and agree to use a reliable method of birth control or remain abstinent duringthe study. Methods of contraception considered acceptable include oral contraceptives, contraceptive patch, intrauterine device, vaginal ring, diaphragm with contraceptive gel, or condom with contraceptive gel

* or are women of non-childbearing potential, defined as: women who have had surgical sterilization (hysterectomy, bilateral oophorectomy, or tubal ligation),
* or women who are ≥ 60 years of age.

Exclusion Criteria:

* Known allergic reactions or hypersensitivity to the active ingredients used or the constituents
* Patients with known skin allergies, multiple drug allergies or multiple allergies to cosmetic products
* Pregnant or breast feeding women
* Patient underwent treatment with any form of head lice treatment within the last 30 days prior to the Screening Visit (day 0)
* Patients with chronic scalp disorder
* Individuals on systemic or topical drugs or medications, including systemic antibiotics, which in the opinion of the investigative personnel may interfere with the study results
* Subjects with hair longer than mid-back
* Patients suspected or known not to follow instructions
* Patients or his/her legal representative who are unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to as a result of their participation in the study
* Previous participation in this study or participation in any other investigational trial within the preceding 30 days
* The patients are investigator site personnel directly affiliated with this study and/or their immediate families. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
* The patients are Oystershell employees or are employees of third-party organizations involved in the study.

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2014-10-13 (Actual); Primary Completion 2015-06-08 (Actual); Study Completion 2015-06-08 (Actual)

PRIMARY OUTCOMES:
Cure Rate superior to 70% for the test product | Day 10
  The primary objective was to show, that the cure rate after local application of Test head lice shampoo is better than a predefined limit. It had to be shown, that the Test head lice shampoo achieved a cure rate superior to 70% (cure rate at the end of day 10, corrected for re-infestation).

SECONDARY OUTCOMES:
Cure Rate superior to 70% for the reference product | Day 10
  The secondary objective was the comparison of the cure rate of the test product with the reference product by using different endpoints. It should be shown that the cure rate on day 10 for the reference product for all baseline infestations is better than the pre-defined limit of 70%.
Superior cure rate to the reference | Day 10
  The secondary objective was the comparison of the cure rate of the test product with the reference product by using different endpoints. It should be shown that the test head lice shampoo has a cure rate superior to the reference.
Non-inferiority rate to the reference | Day 10
  The secondary objective was the comparison of the cure rate of the test product with the reference product by using different endpoints. It should be shown that in case, that superiority could not be shown, the test head lice shampoo is at least not-inferior to the reference. A non-inferiority margin of 7.5% was defined.
Local tolerability | Day 0 (at start and after treatment), Day 1, Day 7 (at start and after treatment), Day 10
  Subjective symptoms (burning, paraesthesia, pruritus) after administration of the investigational products were rated by the patients on a 4-category scale on day 0 and day 7 (0h, 1h p.a.) directly after study drug application as well as on day 1 and day 10 p.a.:
  Score 1 = no Score 2 = mild Score 3 = moderate Score 4 = severe
Global tolerability | Day 10
  Global tolerability was assessed by blinded study staff and by the patient or his/her guardian at day 10. The study staff performed the rating in each case prior to the assessment by the patient to avoid bias. Afterwards, the patient self-assessed the global tolerability.
  The global tolerability was rated on a 4-category scale with:
  Score 1 = very good Score 2 = good Score 3 = moderate Score 4 = poor
Skin irritation assessment | Day 0 (before, at start and after treatment),Day 1, Day 7 (before, at start and after treatment), Day 10
  To investigate a potential irritation of the eyes due to the treatment, the trained and blinded study staff assessed the severity of redness of both eyes within 1 hour before first treatment (baseline), as well as directly after study drug application and after the end of treatment on study day 0, day 1, day 7 (pre-treatment, 0h and 1h p.a.) and on day 10.
  For the assessment of eyes the following 4-category scale as mentioned above were used.
  Score 1 = no Score 2 = mild Score 3 = moderate Score 4 = severe
Eye irritation assessment | Day 0 (before, at start and after treatment),Day 1, Day 7 (before, at start and after treatment), Day 10
  Skin irritation (secondary infection, erythema, excoriation) was assessed by blinded and trained study staff within 1 hour before first treatment (baseline), as well as directly after study drug application and after the end of treatment on study day 0, day 1, day 7 (pre-treatment, 0h and 1h p.a.) and on day 10 .
  For the assessment of skin irritation the following 4-category scale as mentioned above were used.
  Score 1 = no Score 2 = mild Score 3 = moderate Score 4 = severe
Esthetical effect of the anti-lice products | Day 0 (after treatment); day 7 (after treatment)
  The esthetical properties of the investigational products were evaluated to determine the satisfaction by the patients with the product after application using a questionnaire about hair and scalp feeling, greasiness, hair look, shininess and volume. The questioning was performed on day 0 and day 7 after treatment and drying the hair.
  Six questions al with Score 1-4:
  Score 1 = strongly agree Score 2 = agree Score 3 = disagree Score 4 = strongly disagree
Adverse Events (AEs) | Day 0 (at start and after treatment),Day 1, Day 7 (at start and after treatment), Day 10
  An Adverse Event (AE) is any unintended or unfavourable sign (including an abnormal finding), symptom or disease occurring in a subject after signing the informed consent until the last study visit, whether or not the event is believed to be causally related to study medication (IMP) or comparative compound. This definition includes any worsening of conditions that were present at the time of entry into the study (signing of the informedconsent) (see International Conference on Harmonization (ICH-E2A). AEs occurring after signing the informed consent but before administration of study medication are defined as non-treatment-emergent events. Those events are evaluated separately because in these cases a causal relationship with the study medication can be excluded.

OTHER OUTCOMES:
Severity of the lice infestation | Day 0 (before and after treatment),Day 1, Day 7 (before and after treatment), Day 10
  The severity of head lice infestation was judged on a 4-point severity scale:
  * 0 = no relevant infestation (0-4 lice and/or nymph present);
  * 1 = mild (5-9 lice and/or nymphs present);
  * 2 = moderate (10-24 lice and/or nymphs present);
  * 3 = severe (≥ 25 lice and/or nymphs present)

CONTACTS AND LOCATIONS:
Overall Officials: Dörte Wolf, PhD, Principal Investigator — CardioSec Clinical Research GmbH
Locations (1):
- CardioSec Clinical Research GmbH, Erfurt, Germany

IPD SHARING:
Plan to Share IPD: Undecided